CLINICAL TRIAL: NCT00131079
Title: Multi-center Evaluation of the Experimental Program for Physical Activity Promotion (PEPAF), Carried Out by Family Physicians
Brief Title: PEPAF: Evaluation of Family Physician's Effectiveness for Physical Activity Promotion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Collaborators: Preventive Services and Health Promotion Research Network (Other); Castilla-León Health Service (Other); Health Service of Andalucia (Other Government); Castilla-La Mancha Health Service (Other); Dalt Sant Joan primary care center (Health Service of Islas Baleares) (Unknown); Public Health Service of Madrid (Other); Public Health Service of Galicia (Other); Public Health Service of Cataluña (Other); Carlos III Health Institute (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PI020015-G03/170; PI020015; G03/170
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2007-10

CONDITIONS: Exercise; Physical Fitness; Quality of Life
Keywords: Primary Health Care; Physicians, Family; Family Practice; Health Promotion; Randomized Controlled Trials; Multicenter Studies; Physical Fitness; Quality of Life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEPAF (Experimental): General Practitioner's assessment of physical activity level and minimal advice in routine clinical practice supplemented by physical activity prescription to those who accepted an additional 15 minutes appointment.
  Interventions: Behavioral: Experimental Programme for Physical Activity Promotion
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Experimental Programme for Physical Activity Promotion — General practitioner's (GP) physical activity (PA) assessment and advise using a web-based software that prompted open questions to elicit believes about benefits of PA, graphical information about risks of inactivity and examples of type sentences to provide medical advise.
  Educational materials summarizing benefits, risks and motivation.
  Prescription: 15 minutes educational session in which GP negotiated a goal, addressed possible barriers and anticipated solutions using web-based tools for lack of time, community resources, and health problems. Finally, they designed a 3-month PA activity plan that derived in a standardized printed prescription of frequency, duration, intensity and progression of a selected PA or exercise that included a self-monitoring log.
  Arms: PEPAF
Behavioral: Control — Control general practitioners assessed physical activity and performed recruitment in a similar way but offered usual care
  Arms: Control

SUMMARY:
The potential health gains from active lifestyles are very well-known and it is recommended that all adults dedicate at least 30 minutes to activities of at least moderate intensity at least five days a week. What is still not known is how to help sedentary people follow this recommendation, by means of brief interventions feasible in routine general practice. This multi-center study was designed to evaluate the effectiveness of a physical activity promotion program (called PEPAF) implemented in 56 general practices of the Spanish public primary health care system. The study will test the capacity of the program to increase the physical activity level, physical fitness and health related quality of life of sedentary people.

DETAILED DESCRIPTION:
Despite sedentary behavior being one of the strongest risk factors for chronic diseases and mortality, most of the population remains sedentary and evidence is inconclusive that counseling adults in the primary care setting to increase physical activity is effective.

The OBJECTIVE of this randomized clinical trial was to evaluate the effectiveness of an innovative programme to promote physical activity (called PEPAF) implemented by family doctors into daily routine practice. Doctors randomly allocated to the PEPAF group identified sedentary people who visited them for any reason, diagnosed their stage of change and prescribed a written plan of physical activity with those patients ready to change. Those not prepared to change were briefly counseled and given printed materials to motivate them. Patients with cardiovascular disease or other problems meaning that exercise could cause adverse effects were excluded.

Participating people will be followed for 24 months to measure the increase in the level of physical activity from baseline measurement to 6, 12 and 24 months, using 7-day physical activity recall. Health-related quality of life and cardiorespiratory fitness (submaximal cycle ergometer test) will also be measured.

People assigned to the PEPAF group will be COMPARED to patients of family doctors randomly assigned to the control group in which any systematic intervention on physical activity promotion has been postponed until year 2006, except for those patients whose health problems were directly related to a sedentary lifestyle. The average changes observed in the two groups will be compared, on the basis of intention to treat through analysis of covariance. The investigators will use mixed-effect models to take into account intra-patient, intra-doctor and intra-center correlation.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary people who visit the general practitioner for any reason (those who do not dedicate at least 30 minutes to activities of at least moderate intensity at least five days a week).

Exclusion Criteria:

* Disorders of the cardiovascular system
* Transplant recipients
* Renal or hepatic failure
* Severe chronic obstructive pulmonary disease
* Severe mental disorders
* Chronic and acute severe infections
* Metabolic uncontrolled disorders
* Restrictive pathology of muscles, bones and joints
* Complicated pregnancy
* Contact difficulties

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4317 (Actual)
Dates: Start 2003-10; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Physical activity level (7-day Physical Activity Recall [PAR]) | six months from the start of the intervention

SECONDARY OUTCOMES:
Cardiorespiratory fitness | six months from the start of the intervention
Health related quality of life (SF-36) | six months from the start of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Grandes, Dr., Principal Investigator — Primary Care Research Unit of Bizkaia (Basque Health Service)

REFERENCES:
- [Background] Grandes G, Sanchez A, Torcal J, Ortega Sanchez-Pinilla R, Lizarraga K, Serra J; Grupo PEPAF. [Protocol for the multi-centre evaluation of the Experimental Programme Promotion of Physical Activity (PEPAF)]. Aten Primaria. 2003 Nov 15;32(8):475-80. doi: 10.1016/s0212-6567(03)79318-4. Spanish. PMID 14636505
- [Background] Hillsdon M, Foster C, Thorogood M. Interventions for promoting physical activity. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003180. doi: 10.1002/14651858.CD003180.pub2. PMID 15674903
- [Background] Eden KB, Orleans CT, Mulrow CD, Pender NJ, Teutsch SM. Does counseling by clinicians improve physical activity? A summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2002 Aug 6;137(3):208-15. doi: 10.7326/0003-4819-137-3-200208060-00015. PMID 12160371
- [Background] Lopez-de-Munain J, Torcal J, Lopez V, Garay J. Prevention in routine general practice: activity patterns and potential promoting factors. Prev Med. 2001 Jan;32(1):13-22. doi: 10.1006/pmed.2000.0777. PMID 11162322
- [Background] U. S. Department of Health and Human Services. Physical Activity and Health: a report of the Surgeon General. Atlanta, GA: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, National Center for Chronic Disease Prevention and Health Promotion, 1996.
- [Background] Grandes G, Cortada JM, Arrazola A, Laka JP. Predictors of long-term outcome of a smoking cessation programme in primary care. Br J Gen Pract. 2003 Feb;53(487):101-7. PMID 12817354
- [Background] Grandes G, Cortada JM, Arrazola A. An evidence-based programme for smoking cessation: effectiveness in routine general practice. Br J Gen Pract. 2000 Oct;50(459):803-7. PMID 11127170
- [Derived] Grandes G, Sanchez A, Montoya I, Ortega Sanchez-Pinilla R, Torcal J; PEPAF Group. Two-year longitudinal analysis of a cluster randomized trial of physical activity promotion by general practitioners. PLoS One. 2011 Mar 29;6(3):e18363. doi: 10.1371/journal.pone.0018363. PMID 21479243
- [Derived] Grandes G, Sanchez A, Sanchez-Pinilla RO, Torcal J, Montoya I, Lizarraga K, Serra J; PEPAF Group. Effectiveness of physical activity advice and prescription by physicians in routine primary care: a cluster randomized trial. Arch Intern Med. 2009 Apr 13;169(7):694-701. doi: 10.1001/archinternmed.2009.23. PMID 19364999